CLINICAL TRIAL: NCT04597814
Title: The Relationship Between the Tumor Markers and Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: yilunshen2020145
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: the Relationship Between the Tumor Markers and Interstitial Lung Disease Patients
Keywords: carcinoembryonic antigen; carbohydrate antigen 19-9; carbohydrate antigen 125

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — lung specimen after lung transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interstitial lung disease patients: interstitial lung disease patients who need lung transplantation
  Interventions: Other: No Intervention
- non- interstitial lung disease patients: non- interstitial lung disease patients who need thoracic surgery to remove pneumatocele
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The serum levels of carcinoembryonic antigen (CEA), carbohydrate antigen 19-9 (CA19-9), CA125 are often increased in interstitial lung disease patients.

This study was undertaken to investigate the source of these serum tumor markers.

DETAILED DESCRIPTION:
The serum levels of carcinoembryonic antigen (CEA), carbohydrate antigen 19-9 (CA19-9), CA125 are often increased in interstitial lung disease patients.

This study was undertaken to investigate the source of these serum tumor markers.We hypothesis that these tumor markers are released from the lung.

The broncholveolr lvge fluid levels of carcinoembryonic antigen (CEA), carbohydrate antigen 19-9 (CA19-9), CA125 were measured in the interstitial lung disease patients before lung transplantation. The immunohistochemical test was performed in the specimen lung after lung transplantation.

ELIGIBILITY:
Inclusion Criteria

1.Interstitial lung disease patients for lung transplantation

-

Exclusion Criteria:

1. tumor
2. Interstitial lung disease patients could not be performed by lung transplantation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung disease patients for lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
serum levels of carcinoembryonic antigen (CEA) | 6months
  serum levels of carcinoembryonic antigen (CEA)
serum levels of carbohydrate antigen 19-9 (CA19-9) | 6months
  serum levels of carbohydrate antigen 19-9 (CA19-9)
serum levels of carbohydrate antigen 125(CA125) | 6months
  serum levels of carbohydrate antigen 125(CA125)
The alveolar lavage fluid levels of carcinoembryonic antigen (CEA) | 1 week
  The alveolar lavage fluid levels of carcinoembryonic antigen (CEA)
The alveolar lavage fluid levels of carbohydrate antigen 19-9 (CA19-9) | 1 week
  The alveolar lavage fluid levels of carbohydrate antigen 19-9 (CA19-9)
The alveolar lavage fluid levels of carbohydrate antigen 125 | 1 week
  The alveolar lavage fluid levels of carbohydrate antigen 125
The lung tissue levels of carcinoembryonic antigen (CEA) | 1 week
  The lung tissue levels of carcinoembryonic antigen (CEA)
The lung tissue levels of carbohydrate antigen 19-9 (CA19-9) | 1 week
  The lung tissue levels of carbohydrate antigen 19-9 (CA19-9)
The lung tissue levels of carbohydrate antigen 125 | 1 week
  The lung tissue levels of carbohydrate antigen 125

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided